CLINICAL TRIAL: NCT06380257
Title: Anorexia Nervosa and Brain in Adolescence
Status: Not yet recruiting | Type: Observational
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Principal Investigator, Virve Kekkonen, Specialist in adolescent psychiatry, clinical lecturer, Kuopio University Hospital
Other Study IDs: ANBA
Record Dates: First submitted 2024-04-05; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Adolescents diagnosed with anorexia nervosa or atypical anorexia nervosa.
  Interventions: Other: Observational study methods
- Control Group: Healthy adolescents.
  Interventions: Other: Observational study methods

INTERVENTIONS:
Other: Observational study methods — Neuroimaging, body compostion, laboratory tests and psychiatric interview in study and in control groups.

SUMMARY:
Aims of this follow-up study are to investigate effects of anorexia nervosa on brain structure and functions in adolescence.

DETAILED DESCRIPTION:
Anorexia nervosa is severe mental health problem with increased incidence rates in adolescence. Etiology of anorexia nervosa is still mostly unkonwn. Adolescence is also critical period of brain development.

Aims of this follow-up study are to investigate effects of anorexia nervosa on brain structure and functions in both acute and remission state of anorexia nervosa in adolescence.

Study group are young anorexia nervosa patients, and control group are healthy same-aged students.

Research methods include non-invasive brain imaging methods such as Transcranial Magnetic Stimulation (TMS), and Magnetic Resonance Imaging (MRI). Other research methods are assessment of body composition, laboratory tests, self-rated questionnaires and psychiatric interview.

ELIGIBILITY:
Inclusion Criteria:

Study group: 1) age 16-19 years, 2) BMI below 17.5, 3) diagnosis: anorexia nervosa or atypical anorexia nervosa 4) diagnosed within last two years. Inclusion criteria.

Control group : 1) age 16-19 years, 2) BMI over 19.0, 3) No lifetime obesity (BMI over 30) nor eating disorder.

Exclusion Criteria:

1) glucose metabolism disorder or any chronic medical disorder, or medicine with possible effects on neurotransmitters, 2) previous mental health problem (excluded anorexia nervosa or atypical anorexia nervosa in study group), 3) smoking, nicotine products, alcohol or any other substance abuse or dependence, 4) contraindication for used brain imaging method.

Ages: 16 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Target study population is 50 participants. Study group (25 participants) are recruited from North Savo wellbeing services, Adolescent psychiatry outpatient clinic. Control group (25 participants) are recruited from Kuopio restrict lower and upper secondary schools.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2030-08 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Neuroimaging | Baseline and at 3 years' follow-up
  Transcranial magnetic stimulation (TMS) combined with electroencephalogram (EEG)

SECONDARY OUTCOMES:
Neuroimaging | Baseline and at 3 years' follow-up
  Magnetic resonance imaging (MRI)

OTHER OUTCOMES:
Psychiatric evaluation | Baseline and at 3 years' follow-up
  Self-rated questionnaires measuring somatic and mentalh health (such as EDE-Q, BDI, substance use measurements) and structured psychiatric diagnostic interview (SCID)
Body composition measurement | Baseline and at 3 years' follow-up
  InBody body composition measurement (non-invasive method to measure information about the quantity and segmentation of muscle, bone and fat tissue in body and about your basal metabolic rate)
Laboratory tests | Baseline and at 3 years' follow-up
  Blood sample (markers describing undernourishment, more precise description before study)

CONTACTS AND LOCATIONS:
Overall Officials: Virve Kekkonen, M.D., Principal Investigator — Kuopio University Hospital

IPD SHARING:
Plan to Share IPD: Undecided